CLINICAL TRIAL: NCT07197229
Title: Evaluation of Three Months Combined Hospital and Home-Based Tailored Rehabilitation Program in COPD Patients Recently Admitted to Chest Department of Assiut University Hospital
Brief Title: Hospital- and Home-Based Structured Pulmonary Rehabilitation in Recently Admitted COPD Patients: A Quasi-Experimental Study at Assiut University
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Taghreed Essam, resident at the chest department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Combined Pulmonary Rehabilitat
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: ince this is a quasi-experimental single-arm study, there is only one intervention group the Pulmonary Rehabilitation Group: Participants undergo a 12-week structured PR program including both hospital-based sessions (education, structured exercise, nutrition counseling, smoking cessation) and home-based exercises (daily walking, strength training progression).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients diagnosed with moderate-to-severe COPD (confirmed by spirometry) who are clinically stable (Experimental): Participants undergo a 12-week structured PR program including both hospital-based sessions (education, structured exercise, nutrition counseling, smoking cessation) and home-based exercises (daily walking, strength training progression).
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — A tailored pulmonary rehabilitation program combining hospital-based and home-based components over 12 weeksParticipants undergo a 12-week structured PR program including both hospital-based sessions (education, structured exercise, nutrition counseling, smoking cessation) and home-based exercises (daily walking, strength training progression

SUMMARY:
This study evaluates the effect of a structured three-month pulmonary rehabilitation (PR) program, delivered both in-hospital and at home, on exercise capacity, respiratory symptoms, and functional status in stable COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a leading cause of mortality and morbidity worldwide, significantly reducing patients' physical activity and quality of life. This study investigates a tailored pulmonary rehabilitation program combining hospital-based and home-based components over 12 weeks. The hospital component includes patient education, nutritional support, structured exercise training for both upper and lower limbs, and smoking cessation strategies. The home program emphasizes continuity with daily walking, strength exercises, and lifestyle modifications. The program aims to improve exercise capacity, dyspnea scores, and quality of life. Assessments include the six-minute walk test (6MWT), CAT score, mMRC dyspnea scale, spirometry, arterial blood gas analysis, and the St George's Respiratory Questionnaire. Measurements are collected at baseline and after program completion to assess improvements.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD patients diagnosed based on spirometry (post-bronchodilator FEV1/FVC <70%)

Age > 40 years

Moderate to severe COPD stage

Able and willing to participate in rehabilitation program

Exclusion Criteria:

* Age < 40 years

Current acute COPD exacerbation at enrollment

Significant comorbid conditions limiting participation (e.g., uncontrolled diabetes mellitus, uncontrolled hypertension, left-sided heart failure, renal failure, liver cell failure)

Neuromuscular diseases, severe cognitive impairment, or psychiatric disturbance

Pregnant patients

Unwilling to participate in the rehabilitation program

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) | 12 weeks
  Measures the distance (in meters) a patient can walk in six minutes as a marker of exercise capacity and functional endurance.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold MT, Dolezal BA, Cooper CB. Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease: Highly Effective but Often Overlooked. Tuberc Respir Dis (Seoul). 2020 Oct;83(4):257-267. doi: 10.4046/trd.2020.0064. Epub 2020 Aug 10. PMID 32773722